CLINICAL TRIAL: NCT00513565
Title: A Randomised, Placebo-controlled, Double-dummy, Crossover Design Study to Investigate the Changes of fMRI BOLD Activation Induced by Emotional Activation Paradigms Following Single Doses of GSK561679 and Lorazepam (Comparator) in Healthy Subjects
Brief Title: A Study To Investigate Effects Of GSK561679 On Brain Activation During Emotional Processing In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CRS105510
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: GSK561679,; single,; dose,; lorazepam,; fMRI,; BOLD,; healthy volunteers
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo arm (Placebo Comparator): There are single dose treatment arms of GSK561679, lorazepam as well as placebo.
  Interventions: Drug: single dose
- GSK561679 arm (Experimental): There are single dose treatment arms of GSK561679, lorazepam as well as placebo.
  Interventions: Drug: single dose
- lorazepam arm (Active Comparator): There are single dose treatment arms of GSK561679, lorazepam as well as placebo.
  Interventions: Drug: single dose

INTERVENTIONS:
Drug: single dose — Subjects will receive single doses of GSK561679, lorazepam, or placebo at each treatment session.

SUMMARY:
This study will be conducted in healthy volunteers to investigate the effect of single dose GSK561679 on the changes of brain activation, as it compares to an active comparator, lorazepam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Non-smokers
* Body weight 50 kg (110 lbs) or higher, and BMI within the range 19-29.9 kg/m2
* Normal ECG.

Exclusion Criteria:

* Any serious medical disorder or condition.
* Any history of an endocrine disorder.
* Any clinically significant laboratory abnormality.
* History of psychiatric illness.
* Any history of suicidal attempts or behavior.
* History or current diagnosis of acute narrow angle glaucoma.
* Left handed

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09-13 (Actual); Primary Completion 2009-05-14 (Actual); Study Completion 2009-05-14 (Actual)

PRIMARY OUTCOMES:
Differences in fMRI brain activation (BOLD) response in specific brain regions | conducted the duration of the study

SECONDARY OUTCOMES:
Physiologic changes | during & after fMRI session
Visual Analogue Scale measurement of physical reactions | duration of study
Blood level of GSK561679 | collected during fMRI session
Vital signs & ECG recording | duration of the study
Lab tests for blood & urine | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, La Jolla, California, United States

REFERENCES:
- See also: Results for study CRS105510 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CRS105510?search=study&study_ids=CRS105510#rs